CLINICAL TRIAL: NCT03374709
Title: Pilot Study of Oxtellar XR (Oxcarbazepine Extended Release) in Neurology Patients With Trigeminal Neuralgia
Brief Title: Oxtellar Extended Release (Oxcarbazepine Extended Release) Patients With Trigeminal Neuralgia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Resource and time constraints were encountered by product manufacturer and study team.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-1398
Record Dates: First submitted 2017-08-09; First posted 2017-12-15 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): This arm includes subjects who have been prescribed Oxtellar XR 150Mg Extended Release Tablets.
  Interventions: Drug: Oxtellar XR 150Mg Extended Release Tablet

INTERVENTIONS:
Drug: Oxtellar XR 150Mg Extended Release Tablet — Oxtellar XR
  Other Names: Oxtellar XR 300Mg Extended Release Tablet; Oxtellar XR 600Mg Extended Release Tablet

SUMMARY:
To evaluate the affect Oxtellar XR (Extended Release) has on neurology patients with trigeminal neuralgia (TN), and if it impacts their quality of life.

DETAILED DESCRIPTION:
Oxcarbazepine has been used off-label for TN for many years, but has a twice daily dosing. With the once daily dosing it should theoretically help with patient adherence and possibly decrease side effects, which is common with extended release formulations. Specifically the investigators are looking at how well tolerated Oxtellar XR is, and if it has the same efficacy as standard treatments. It is a pilot study, so it will be difficult to gather data and have powerful outcomes, but this will give pilot data for future trials. Patients will be screened for inclusion and exclusion criteria and after will participate in 3 visits following the initial one. Various tests will be administered to measure treatment satisfaction and tolerability throughout the visits. The patients will not have to pay for any of the study visits or medications. A parking voucher will be provided as needed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 to 75
* Subject reported history of trigeminal neuralgia average pain rated as > lower end of moderate on the VAS
* Trigeminal neuralgia diagnosis (Primary or type 1 or Idiopathic TN)
* History of pain rated as at least a 4 on the visual analog scale (VAS)
* Treatment naïve
* Patients who do not tolerate carbamazepine
* Women of reproductive age who agree to highly effective birth control
* Complete Blood Count (CBC) 30 days prior to entering study
* Comprehensive metabolic panel (CMP) 30 days prior to entering study

Exclusion Criteria:

* Intolerance/Hypersensitivity to Trileptal, Oxcarbazepine, or Oxtellar
* Psychosis, drug/alcohol misuse, or malignancy (except skin cancer) within the last 2 years
* Any clinically significant medical condition that would prevent study from being completed safely (determined by subjects current neurologist)
* Current seizure disorder or history of seizures
* Pregnant females
* Breastfeeding females
* Women of reproductive age not using or unwilling to utilize highly effective contraception (defined as double-barrier method)
* A severe pain condition, other than trigeminal neuralgia, which may impair the self-assessment of pain due to trigeminal neuralgia
* Concurrent medication treatment with: Equetro, Phenytoin, Dilantin, Phenytek, Oxcarbazepine, Trileptal, Rifampin, Rifadin, Rimactane and St. John Wort
* Renal impairment or hemodialysis
* Hepatic impairment
* History of hyponatremia (serum sodium < 125 ng/dL)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Change in pain associated with trigeminal neuralgia (BPI) | Weeks 2, 6, and 10 following screening
  Pain associated with trigeminal neuralgia as measured by the Brief Pain Inventory (BPI) facial.
Change in pain associated with trigeminal neuralgia (VAS) | Weeks 2, 6, and 10 following screening
  Pain associated with trigeminal neuralgia as measured by a Visiual Analog Scale (VAS).

SECONDARY OUTCOMES:
Change in Quality of Life | Weeks 2, 6, and 10 following screening
  The Subjects Quality of life will be evaluated based on the their responses to the following endpoint: treatment satisfaction QOL questionnaire
Change in Safety: Number of Attacks | Weeks 2, 6, and 10 following screening
  The subjects Safety profile will be measured based upon the number of attacks experienced.
Change in Safety: SF-12 Survey | Weeks 2, 6, and 10 following screening
  The subjects Safety profile will be measured based upon completion of the SF-12 survey
Change in Safety: Heart Rate | Weeks 2, 6, and 10 following screening
  The subjects Safety profile will be measured based upon any noted changes in heart rate.
Change in Safety: Blood Pressure | Weeks 2, 6, and 10 following screening
  The subjects Safety profile will be measured based upon any noted changes in Blood pressure.
Change in Safety: CBC | Weeks 2, 6, and 10 following screening
  The subjects Safety profile will be measured based upon a complete blood count (CBC).
Change in Safety: CMP | Weeks 2, 6, and 10 following screening
  The subjects Safety profile will be measured based upon a Comprehensive Metabolic Panel (CMP).
Change in Treatment Satisfaction | Weeks 2, 6, and 10 following screening
  Treatment satisfaction will be measured through the completion of the Treatment Satisfaction Questionnaire For Medication (TSQM).
Change in Tolerability: Number of Attacks | Weeks 2, 6, and 10 following screening
  Change in Tolerability will be measured by the number of attacks.
Change in Tolerability: SF-12 Survey | Weeks 2, 6, and 10 following screening
  Change in Tolerability will be measured by the completion of the SF-12 survey.
Change in Tolerability: Vital Signs | Weeks 2, 6, and 10 following screening
  Change in Tolerability will be measured by vital signs.
Change in Tolerability: CBC | Weeks 2, 6, and 10 following screening
  Change in Tolerability will be measured by a complete blood count (CBC).
Change in Tolerability: CMP | Weeks 2, 6, and 10 following screening
  Change in Tolerability will be measured by a comprehensive metabolic panel (CMP).
Change in Tolerability: TSQM | Weeks 2, 6, and 10 following screening
  Change in Tolerability will be measured by the completion of the Treatment Satisfaction Questionnaire For Medication (TSQM).

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Bainbridge, PharmD, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Background] Available at: http://trigeminalneuralgia-ronaldbrismanmd.com/Trigeminal-Neuralgia-MS.html. Accessed December 12, 2016.
- [Background] Available at: http://fpa-support.org/tn-and-ms-2/. Accessed December 12, 2016
- [Background] Cruccu G, Finnerup NB, Jensen TS, Scholz J, Sindou M, Svensson P, Treede RD, Zakrzewska JM, Nurmikko T. Trigeminal neuralgia: New classification and diagnostic grading for practice and research. Neurology. 2016 Jul 12;87(2):220-8. doi: 10.1212/WNL.0000000000002840. Epub 2016 Jun 15. PMID 27306631
- [Background] Cruccu G, Gronseth G, Alksne J, Argoff C, Brainin M, Burchiel K, Nurmikko T, Zakrzewska JM; American Academy of Neurology Society; European Federation of Neurological Society. AAN-EFNS guidelines on trigeminal neuralgia management. Eur J Neurol. 2008 Oct;15(10):1013-28. doi: 10.1111/j.1468-1331.2008.02185.x. Epub 2008 Aug 21. PMID 18721143
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Chen HI, Lee JY. The measurement of pain in patients with trigeminal neuralgia. Clin Neurosurg. 2010;57:129-33. No abstract available. PMID 21280505
- [Background] Available at: http://www.quintiles.com/landing-pages/treatment-satisfaction-questionnaire-for-medication-tsqm. Accessed December 12, 2016
- [Background] Sandhu SK, Halpern CH, Vakhshori V, Mirsaeedi-Farahani K, Farrar JT, Lee JY. Brief pain inventory--facial minimum clinically important difference. J Neurosurg. 2015 Jan;122(1):180-90. doi: 10.3171/2014.8.JNS132547. PMID 25361481